CLINICAL TRIAL: NCT05555381
Title: Anxiety, Stress and Sleep Problems in People With Early Onset Dementia
Acronym: Young-D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Collaborators: Odisee University college for applied sciences (Other)
Responsible Party: Principal Investigator, Julie Vanderlinden, Principal investigator, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Young-D
Record Dates: First submitted 2022-06-02; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Early Onset Dementia; Young Onset Dementia; Stress; Distress, Emotional; Anxiety; Sleep Problem; Sleep; Insomnia
MeSH Terms: conditions — Anxiety Disorders; Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (pilot study) (Experimental): * needs detection by means of survey and interviews (mixed-methods)
  * 6 week program (1 hour) on a weekly basis including cognitive behavioural therapy, sleep/stress hygiene education, heart coherence exercises, mindfulness and relaxation exercises
  Interventions: Behavioral: young-D program

INTERVENTIONS:
Behavioral: young-D program — * needs detection by means of survey and interviews (mixed-methods)
  * 6 week program (1 hour) on a weekly basis including cognitive behavioural therapy, sleep/stress hygiene education, heart coherence exercises, mindfulness and relaxation exercises

SUMMARY:
The aim of this study is to

* detect and assess needs of people with early onset dementia regarding anxiety, stress and sleep
* implement a 6 week intervention pilot study in wich weekly (hourly) sessions are implemented in day care settings in order to decrease anxiety, stress and sleep problems in people with early onset dementia

DETAILED DESCRIPTION:
1. needs detection by means of survey and interviews
2. implementation of a 6 week program in day care facilities

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with early onset dementia before age of 65Y

Exclusion Criteria:

* severe dementia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
anxiety (GAD7 validated questionnaire) | 6 weeks
  this is a subjective survey that measures the level of anxiety in daily life. It is a score of 7 items with a min of 0 and a max of 21. A higher score indicates a higher anxiety.
stress (perceived stress scale, PSS, validated questionnaire) | 6 weeks
  this is a subjective survey that measures the level of stress in daily life. It is a score of 10 items with a min of 0 and a max of 40. A higher score indicates a higher stress level.
sleep (Insomnia severity index, ISI, validated questionnaire) | 6 weeks
  this is a subjective survey that measures the level of insomnia. It is a score of 7 items with a min of 0 and a max of 28. A higher score indicates a worse level of insomnia
sleep (actigraph) | 6 weeks
  this is an objective measurement that measures the sleep quantity

SECONDARY OUTCOMES:
emotional well being (WEMWBS, Warwick emotional mental wellbeing scale) | 6 weeks
  this is a subjective survey that measures the level of emotional well being in daily life. It is a score of14 items with a min of 0 and a max of 77. A higher score indicates a better wellbeing.
quality of life (QoL) (quality of life in dementia, QUALIDEM) | 6 weeks
  this is a subjective survey that measures the level of QoL in daily life. It is a score of 40 items with a min of 0 and a max of 160. Per (7) subscales the scores are cumulated.
heart rate variance (HRV) | 6 weeks
  this is an objective measurement that measures level of HRV in daily life, using (non-invasive photoplethysmography)
Depression (Patient Health Questionnaire PHQ-9, validated questionnaire) | 6 weeks
  this is a subjective survey that measures the level of depression in daily life. It is a score of 10 items with a min of 0 and a max of 27. A higher score indicates a more severe level of depression

CONTACTS AND LOCATIONS:
Overall Officials: Julie Vanderlinden, PhD, Principal Investigator — Odisee University of Applied Sciences
Locations (2):
- Belgium (2):
  - Odisee University of Applied Sciences, Brussel, Flanders
  - Familiezorg Oost Vlaanderen, Ghent, Oost-Vlaanderen